CLINICAL TRIAL: NCT02690675
Title: Iron Supplement Effect Over Immune System and Neurobehavioral Child Development.
Brief Title: Iron Supplement Effect on Child Development
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Rovira i Virgili (Other)
Responsible Party: Principal Investigator, Victoria Arija Val, University Professor, University Rovira i Virgili
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: EC81/00128
Record Dates: First submitted 2016-02-11; First posted 2016-02-24 (Estimated); Last update posted 2016-02-25 (Estimated); Status verified 2016-02

CONDITIONS: Neurodevelopmental Disorders; Lactation
Keywords: Neurodevelopment; Bayley Scale; Growth; Iron fortification
MeSH Terms: conditions — Neurodevelopmental Disorders; Breast Feeding

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention high-iron fortified milk (Experimental): This group received a high dose of iron by formula milk (1.2mg/100mL) between 6 and 12 months of age.
  Interventions: Dietary Supplement: Iron fortified formula milk
- Intervention low-iron fortified milk (Experimental): This group received a low dose of iron by formula milk (0.4mg/100mL) between 6 and 12 months of age.
  Interventions: Dietary Supplement: Iron fortified formula milk

INTERVENTIONS:
Dietary Supplement: Iron fortified formula milk — One group received formula milk fortified with 1.2 mg/100 mL and the other group 0.4 mg/100mL between 6 and 12 months of age.

SUMMARY:
Objective: To evaluate the effect of Iron supplement with two different amounts (one in the higher limit and another in the lower limit of the suggested amount) according to the presence of mutations in the HFE gene in the physical, immune and neurobehavioral development in the 6 to 12 moth toddlers.

Methodology: Subjects: 340 toddlers coming from Paediatric Serves of Sant Joan Hospital. Methods: At 6 and 12 months it done clinical history, food registry, biochemist determinations: haemoglobin, iron, transferrin, ferritin, reactive C protein and immune response (IL4, IL10, IL6 IFN, IgA, IgM, IgG, IgE). Mutations in the HFE gene: C282Y, H63D, S65D and hepcidin gene. Mental, psychomotor and behavioual development (Bayley Scales of Infant Development 2on Edition: 1993). We evaluate the level of language and communication (MacArthur), regulation and sensory process (Infant Toddler Symptom Checklist), familiar and environment surroundings (Scale Health General Parental Stress Index).

DETAILED DESCRIPTION:
Design: Randomised Clinical Trial with two groups of intervention. Group A received high-iron fortified milk (1.2mg/100mL) and Group B received low-iron fortified milk (0.4mg/100mL).

Inclusion criteria: caucasian new-borns, term infants.

Exclusion criteria:

* Families that refuse enter at the follow-up.
* Low-birth weight or preterm infants.
* Anaemic infants.
* Infants with congenital defects, immunodeficiency or hypothyroidism.
* Infants with diseases that requires intensive care.

ELIGIBILITY:
Inclusion Criteria:

* Caucasian infants
* Healthy term infants

Exclusion Criteria:

* Families that do not understand Spanish or Catalan
* Anaemic infants at birth
* Infants with important diseases

Max Age: 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 133 (Actual)
Dates: Start 2006-05; Primary Completion 2009-06 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Mental and psychomotor development with BSID (Bayley Scale of Infant Development) at 12 months. | 12 months

SECONDARY OUTCOMES:
Height at 12 months measured in centimeters | 12 months
Weight at 12 months measured in grams | 12 months
Head circumference at 12 months measured in centimeters | 12 months
Risk of infections at 12 months measured qualitatively from record of presence or not of various infections as bronchitis, rhinitis, otitis etc. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Victoria Arija Val, Professor, Principal Investigator — University Rovira i Virgili

IPD SHARING:
Plan to Share IPD: Yes
The investigators plan to share data in a submitted article in 2016

REFERENCES:
- [Derived] Iglesias Vazquez L, Canals J, Voltas N, Jardi C, Hernandez C, Bedmar C, Escribano J, Aranda N, Jimenez R, Barroso JM, Ribot B, Arija V. Does the fortified milk with high iron dose improve the neurodevelopment of healthy infants? Randomized controlled trial. BMC Pediatr. 2019 Sep 5;19(1):315. doi: 10.1186/s12887-019-1679-0. PMID 31488098